CLINICAL TRIAL: NCT00520923
Title: A Multi-Center, Inpatient, Phase 2, Double-blind, Placebo-Controlled Dose Ranging Study of LY2140023 in Patients With DSM-IV Schizophrenia
Brief Title: A Study for Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11757; H8Y-MC-HBBI
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): 160mg of LY2140023, taken orally as 80mg twice daily, for up to 4 weeks.
  Interventions: Drug: LY2140023
- 2 (Experimental): 80mg of LY2140023, taken orally as 40mg twice daily, for up to 4 weeks.
  Interventions: Drug: LY2140023
- 3 (Experimental): 40mg of LY2140023, taken orally as 20mg twice daily, for up to 4 weeks.
  Interventions: Drug: LY2140023
- 4 (Experimental): 10mg of LY2140023, taken orally as 5mg twice daily, for up to 4 weeks.
  Interventions: Drug: LY2140023
- 5 (Placebo Comparator): Placebo of LY2140023, taken orally twice daily, for up to 4 weeks.
  Interventions: Drug: Placebo
- 6 (Active Comparator): Placebo, taken orally every morning, followed by Olanzapine 15mg taken orally every evening for up to 4 weeks.
  Interventions: Drug: Olanzapine; Drug: Placebo

INTERVENTIONS:
Drug: LY2140023 — 80mg, PO (by mouth) BID (twice a day) for up to 4 weeks.
  Arms: 1
Drug: LY2140023 — 40mg, PO (by mouth) BID (twice daily) for up to 4 weeks.
  Arms: 2
Drug: LY2140023 — 20mg, PO (by mouth) BID (twice daily) for up to 4 weeks.
  Arms: 3
Drug: LY2140023 — 5mg, PO (by mouth) BID (twice daily) for up to 4 weeks.
  Arms: 4
Drug: Olanzapine — 10mg, PO (by mouth) QPM (every evening) for the first 3 days, then 15mg PO QPM, for up to 4 weeks.
  Arms: 6
Drug: Placebo — Taken PO (by mouth) QAM (every morning) for up to 4 weeks.
  Arms: 6
Drug: Placebo — Taken PO (by mouth) BID (twice daily) for up to 4 weeks.
  Arms: 5

SUMMARY:
The purpose of this study is to test the hypothesis that 1 or more dose levels of LY2140023 given orally to patients with schizophrenia twice daily for 4 weeks will have significantly greater effect than placebo.

ELIGIBILITY:
Some Inclusion Criteria:

* Patients must have a diagnosis of Schizophrenia as defined in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) (Disorganized, 295.10; Catatonic, 295.20; Paranoid, 295.30; Residual, 295.60; or Undifferentiated, 295.90) and confirmed by the Structured Clinical Interview for DSM-IV (SCID).
* Patients must meet the following psychopathologic severity criteria at Visit 1: Brief Psychiatric Rating Scale (BPRS) total score, extracted from the Positive and Negative Syndrome Scale (PANSS), of at least 45 (18-item version, in which 1 indicates "absent" and 7 indicates "severe"). In addition, item scores of at least 4 (moderate) will be required on 2 of the following BPRS items: conceptual disorganization, suspiciousness, hallucinatory behavior, and/or unusual thought content.
* Patients must receive a rating of 4 (moderately ill) or greater on the Clinical Global Impression-Severity (CGI-S) scale at Visit 1.
* Patients in whom, in the opinion of the investigator, a switch to another antipsychotic medication or initiation of an antipsychotic medication is acutely indicated.

Some Exclusion Criteria:

* Patients in whom treatment with olanzapine or placebo is relatively or absolutely clinically contraindicated.
* Patients who have a history of inadequate response to an adequate treatment trial with olanzapine, in the opinion of the investigator.
* Patients who have received treatment with olanzapine within 6 weeks prior to Visit 1.
* Patients who have received treatment with clozapine at doses greater than 200 mg daily within 12 months prior to Visit 1, or who have received any clozapine at all during the month before Visit 1.
* Patients who have a history of an inadequate response, in the opinion of the investigator, to 2 or more adequate antipsychotic medication trials of at least 8 weeks duration in the past 12 months prior to Visit 1.
* Patients with acute, serious, or unstable medical conditions, including (but not limited to) inadequately controlled diabetes (hemoglobin A1c (HbA1c) 8%), severe hypertriglyceridemia (fasting triglycerides 5.6 mmol/L, recent cerebrovascular accidents, serious acute systemic infection or immunologic disease, unstable cardiovascular disorders (including ischemic heart disease), malnutrition, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, or hematologic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) total score | over 4 weeks of treatment

SECONDARY OUTCOMES:
PANSS subscores: positive subscore; negative subscore; general psychopathology subscore and cognitive subscore | over 4 weeks of treatment
Clinical Global Impression-Severity (CGI-S) | over 4 weeks of treatment
Drug Attitude Inventory-10 (DAI-10) | over 4 weeks of treatment
Response and Remission Rates | over 4 weeks of treatment
Assessment of Cognition in Schizophrenia (BACS) Symbol Coding Task | over 4 weeks of treatment
Montgomery-Asberg Depression RatingScale (MADRS) | over 4 weeks of treatment
Safety and Tolerability | over 4 weeks of treatment
Pharmacokinetics | over 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banfield
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lanús Este
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munro
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Croatia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Split
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aachen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Portugal (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khot'kovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lipetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Samara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Village Nikolskoe
- South Africa (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johannesburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Randburg

REFERENCES:
- [Derived] Kinon BJ, Millen BA, Zhang L, McKinzie DL. Exploratory analysis for a targeted patient population responsive to the metabotropic glutamate 2/3 receptor agonist pomaglumetad methionil in schizophrenia. Biol Psychiatry. 2015 Dec 1;78(11):754-62. doi: 10.1016/j.biopsych.2015.03.016. Epub 2015 Mar 19. PMID 25890643
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com